CLINICAL TRIAL: NCT02158559
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Trial of the Effect of Danhong Injection on Microcirculation in the Treatment of Patients With STEMI(ST- Elevation Myocardical Infarction) After the PTCA Surgery.
Brief Title: the Effect of Danhong Injection on Microcirculation in the Treatment of Patients With STEMI After the PTCA Surgery.
Acronym: Danhong
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Bozhiyin T&S Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DH-140318-01
Record Dates: First submitted 2014-05-29; First posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — danhong; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Danhong Injection (Experimental): Danhong injection 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 7 days;
  Interventions: Drug: Danhong Injection
- Normal Saline (Placebo Comparator): 0.9% sodium chloride solution 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 7 days;
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Danhong Injection — Danhong injection 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 7 days;
  Arms: Danhong Injection
Drug: Normal Saline — 0.9% sodium chloride solution 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 7 days;
  Arms: Normal Saline

SUMMARY:
This study focused on the effect of Danhong injection on microcirculation in the treatment of patients with STEMI(ST-elevation myocardical infarction) after the PTCA surgery.

DETAILED DESCRIPTION:
Research Topic.

* A randomized, double-blind, placebo-controlled, multi-center clinical trial of the effect of Danhong Injection on microcirculation in the treatment of patients with STEMI(ST- elevation myocardical infarction) after the PTCA surgery.

Research Purpose.

* This study focused on the effect of Danhong injection on microcirculation in the treatment of patients with STEMI(ST-elevation myocardical infarction) after the PTCA surgery.

Research design.

* A randomized, double-blind, placebo-controlled, multi-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite or laboratory-supported diagnosis of STEMI ,with the indication of PTCA surgery.
* 18≤Age≤75;
* Agreed to join in the study and signed the inform consent form.

Exclusion Criteria:

* Cardiogenic shock , Killip III-IV degree , papillary muscle rupture , septal perforation , episodes of ventricular tachycardia and ventricular fibrillation after electrical cardioversion , temporary pacemaker implanted AVB III degree.
* Past history of PCI and CABG
* Acute or chronic infectious diseases(for example severe pneumonia);
* Recent history of hemorrhagic stroke(within six months)
* Combined with liver and kidney dysfunction;
* History of valvular heart disease;
* Congenital heart disease or Pulmonary hypertension;
* All kinds of history of cardiomyopathy;
* Bleeding and other thrombotic diseases;
* Severe anemia , thrombocytopenia , Other diseases of the blood system;
* Cancer , Autoimmune disease , All kinds of the patients who use the glucocorticoid and immunosuppressor;
* Menstrual period women, pregnant women and lactating women, pregnancy test positive or recent family planning.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
After 7 days surgery used magnetic resonance assessed myocardial perfusion and myocardial function. | 1 week